CLINICAL TRIAL: NCT06427200
Title: Efficacy and Safety of Lactoferrin in Heart Failure Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, reham mohamed saied salem, Teaching assistant at Faculty of Pharmacy Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL(3530); IHC00072 (Other: the general organization for teaching hospitals and institutes (GOTHI))
Record Dates: First submitted 2024-05-18; First posted 2024-05-23 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Lactoferrin; oral iron; reduced ejection fraction; iron deficiency; heart failure; clinical trial
MeSH Terms: conditions — Iron Deficiencies; Heart Failure | interventions — Iron; Lactoferrin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group "oral iron" (Experimental)
  Interventions: Drug: oral Iron
- group "lactoferrin" (Experimental)
  Interventions: Drug: Lactoferrin
- group "lactoferrin and oral iron" (Experimental)
  Interventions: Drug: lactoferrin and oral iron

INTERVENTIONS:
Drug: oral Iron — oral iron once daily during or after meals as add-on therapy for 12 weeks.
  Arms: group "oral iron"
Drug: Lactoferrin — lactoferrin twice daily before meals as add-on therapy for 12 weeks.
  Arms: group "lactoferrin"
Drug: lactoferrin and oral iron — lactoferrin twice daily before meals and oral iron once daily during or after meals as add-on therapy for 12 weeks.
  Arms: group "lactoferrin and oral iron"

SUMMARY:
This study will be conducted to determine the efficacy and safety of lactoferrin versus oral iron versus lactoferrin plus oral iron as an add on therapy in reduced ejection fraction heart failure patients with iron deficiency.

•Patients will be randomly distributed into the three groups

* All patients will be subjected to baseline data assessment
* Follow up after 12 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years old.
2. Chronic heart failure (> 6 months duration) with reduced ejection fraction defined as LVEF ≤ 40%.
3. NYHA-class II or III or IV with stable symptoms for at least the past 3 months.
4. Stabilized on beta blockers, renin-angiotensin system inhibitor (ACEI/ARB) or angiotensin receptor-neprilysin inhibitors (ARNIs), mineralocorticoid receptor antagonists (MRAs) and sodium-glucose co-transporter 2 Inhibitors (SGLT2i) and diuretics as needed.
5. No dose changes of heart failure drugs during the last 2 weeks (exception: diuretics)
6. No introduction of a new heart failure drug class during the last 4 weeks.
7. Iron deficiency: serum ferritin level of 15 to 100 ng/mL or a serum ferritin level of 101 to 299 ng/mL with transferrin saturation of less than 20%.

Exclusion Criteria:

* 1. Arrythmia including atrial fibrillation (AF) with poorly controlled ventricular rate at rest (> 100 beats/min).

  2. Recent cardiac related hospitalizations in the past 3 months. 3. Known active infection. 4. Associated chronic medical disorder (chronic kidney disease (creatinine clearance < 60 ml/min), liver disease (ALT or AST > 3× upper limit of normal), peptic ulcer or chronic blood loss).

  5. Associated bleeding disorder. 6. Previous iron supplement in past 3 months. 7. Anemia requiring blood transfusion (haemoglobin (Hb) < 7 g/dL). 8. Folic acid or vitamin B12 deficiency. 9. Hypersensitivity to lactoferrin or iron. 10. Haemoglobinopathies (G6PD, thalassemia's, sickle cell disease). 11. Pregnancy and lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life (HR-QoL) | 3 months
  • Change in health-related quality of life (HR-QoL) as evaluated by Minnesota Living with Heart Failure Questionnaire (MLHFQ) minimum score:0 maximum score:105 minimum score is a better outcome